CLINICAL TRIAL: NCT01575301
Title: DIabetes REsearCh on Patient sTratification (DIRECT): GLP-1R Agonists
Acronym: DIRECTGLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ewan Pearson, Chief Investigator, University of Dundee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011DIRECT01 (GLP)
Record Dates: First submitted 2012-03-29; First posted 2012-04-11 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Diabetes
Keywords: GLP-1R agonist; biomarker
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exenatide; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Exenatide, Liraglutide — Dosage, frequency and duration not specified by protocol
  Other Names: Byetta; Victoza

SUMMARY:
The purpose of this study is to collect a cohort of patients treated with GLP-1R Agonists and to assess phenotypic, genetic and genomic biomarkers of glycaemic response to these agents.

DETAILED DESCRIPTION:
To develop a cohort of patients treated with GLP-1 R Agonists who are phenotyped at baseline and at 6 month follow up to determine clinical, imaging and other biomarker predictors of glycaemic response to GLP-1R Agonists. The hypothesis is that one, or a combination, of these biomarkers is associated with glycaemic response to GLP-1R Agonists. The primary outcome is therefore HbA1c reduction after 6 months of GLP-1R A treatment.

This is a cohort study of 800 patients being treated with either exenatide or liraglutide for 6 months, and carried out in 4 UK centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes where a clinical decision has been made to commence a GLP-1R agonist
* Either:

  1. On any combination of oral hypoglycaemic agents
  2. On Insulin (+/- oral hypoglycaemic agents)
* HbA1c ≥7.5% (58mmol/mol) and HbA1c < 12% (108mmol/mol)
* White European
* Age ≥ 18 and < 80

Exclusion Criteria:

* Type 1 diabetes
* HbA1c <7.5% (58 mmol/mol)
* HbA1c ≥ 12% (108 mmol/mol)
* Pregnancy or lactation
* Any other significant medical reason for exclusion as determined by the investigator
* Inability to consent
* Participating in a CTIMP during the study period and within 30 days prior to study start.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c between baseline and 6 months | 6 months
  The primary outcome is the change in HbA1c (absolute difference between the baseline and 6 month measure) in mmol/mol

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Pearson, Principal Investigator — University of Dundee
Locations (4):
- United Kingdom (4):
  - Ninewells Hospital, Dundee, Angus
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Oxford Hospitals NHS Trust, Oxford, Oxfordshire
  - Newcastle Hospitals NHS Trust, Newcastle, Teeside